CLINICAL TRIAL: NCT02625285
Title: Validation of New G6PD Point of Care Tests (Biosensors) Against Gold Standard Quantitative Spectrophotometry and Genotyping
Brief Title: Validation of New G6PD Point of Care Tests Against Gold Standard Quantitative
Acronym: Biosensors
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: PATH (Other)
Responsible Party: Sponsor
Other Study IDs: SMRU1501
Record Dates: First submitted 2015-12-04; First posted 2015-12-09 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Validation; Biosensors; Genotyping

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Two blood samples will be withdrawn from participants; one sample will be taken by finger-stick (200 µl) and one sample (0.5 ml) will be taken by arm venipuncture. The blood from capillary sample will be used to assess G6PD activity using the POC tests, CBC and laboratory based quantitative tests. The venous blood will be used for reference standard quantitative G6PD assays, Hb typing analysis, CBC and buffy-coat will be stored for DNA extraction for G6PD genotyping only; leftover blood will be discarded.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- G6PD Deficient Volunteers: * Subjects with age ≥ 18 years
  * Male and female
  * Previously tested G6PD deficient at SMRU clinic
- G6PD Intermediate or Heterozygous Volunteers: * Subjects with age ≥ 18 years
  * Female
  * Previously tested G6PD intermediate or heterozygous for G6PD variants at SMRU clinic
- G6PD-Normal Volunteers: * Subjects with age ≥ 18 years
  * Male and female
  * Previously tested G6PD normal at SMRU clinic

SUMMARY:
This is a laboratory research to evaluate performances of quantitative POC G6PD tests (Biosensors) against gold standard quantitative laboratory based tests and genotyping.

DETAILED DESCRIPTION:
Radical cure of P. vivax malaria can be achieved using large doses of primaquine which have shown to cause some degree of hemolysis even in subjects who tested normal by the conventional qualitative G6PD tests. Different regimens of drug might be more appropriate in subjects with intermediate G6PD activity which can be currently measured only in well equipped laboratories. Validation of new qualitative and quantitative point-of-care tests is essential to for safe deployment of standard and new radical cure regimens against Plasmodium vivax.

This study will evaluate performances of quantitative POC G6PD tests (Biosensors) against gold standard quantitative laboratory based tests and genotyping. Patients will be searched from the electronic record database to identify up to 150 patients with the following characteristics: approximately 50 G6PD-deficient men and women (however only a very small percent of deficients are homozygous women) approximately 50 G6PD-heterozygous women with intermediate activity, and approximately 50 G6PD-normal individuals and patients who meet the screening criteria will be contacted at their home by a clinic staff member. The home visitor will explain study details and invite to participate in the study. If the patients express interest in participating, they will be directed to visit the following month at the clinic where they usually receive care.

After signing the informed consent form, two blood samples will be withdrawn; one sample will be taken by finger-stick (200 µl) and one sample (0.5 ml) will be taken by arm venipuncture. The blood from capillary sample will be used to assess G6PD activity using the POC tests, CBC and laboratory based quantitative tests. The venous blood will be used for reference standard quantitative G6PD assays, Hb typing analysis, CBC and buffy-coat will be stored for DNA extraction for G6PD genotyping only; leftover blood will be discarded.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with age ≥ 18 years
* Subjects willing to participate and sign informed consent form
* Male and Female
* Previously tested G6PD deficient, G6PD normal and G6PD intermediate or heterozygous for G6PD variants at SMRU clinic

Exclusion Criteria:

* Patients with severe malaria or other severe or any acute illness
* Patients who received a blood transfusion in the last 3 months
* Patients who received primaquine in the past 1 month (this is to ensure that previous characterization of phenotype in the healthy subject has not been influenced by a recent hemolytic reaction)
* Patients who have not had a critical illness or received other hemolytic drugs (this is to ensure that previous characterization of phenotype in the healthy subject has not been influenced by a recent hemolytic reaction)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The total sample size will be 150 patients, using targeted enrollment to achieve a convenience sample of approximately 50 G6PD deficient volunteers (male and female), approximately 50 G6PD intermediate or heterozygous female volunteers, and the remaining will be G6PD-normal volunteers with a 1:1 male/female ratio.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2017-01-24 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
correlation in G6PD activity | at enrollment
  determined by the Biosensors and the spectrophotometric gold standard.

SECONDARY OUTCOMES:
correlation in Hemoglobin levels | at enrollment
  determined by the Biosensors and the automated blood analyzer.
Determine association between one or more quantitative POC G6PD test (Biosensor) and the flow cytometry-based G6PD test | at enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Shoklo Malaria Research Unit,, Mae Sot, Changwat Tak, Thailand